CLINICAL TRIAL: NCT02088281
Title: Mechanistic Study of Indigo Naturalis in Treating Psoriasis: Local or Systemic Manipulation of Inflammation and Induction of Immunoregulation
Brief Title: Mechanistic Study of Indigo Naturalis in Treating Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSC 101-2320-B-182-021-MY3
Record Dates: First submitted 2012-12-10; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2012-10

CONDITIONS: Psoriasis Vulgaris
Keywords: Indigo naturalis, indirubin, Th1 cells, Th17 cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indigo naturalis extract in oil ointment (Experimental): Indigo naturalis extract in oil ointment: each gram of ointment contains 200 μg±20 μg of indirubin.
  Interventions: Drug: Indigo naturalis extract in oil ointment

INTERVENTIONS:
Drug: Indigo naturalis extract in oil ointment — Apply 0.5 g of INEO ointment per 10 x 10 cm psoriasis lesion twice daily.
  Other Names: INEO ointment

SUMMARY:
The potential effect of indigo naturalis on the immune system is unknown. The investigators hypothesize that the therapeutic effect of indigo naturalis in psoriasis may involve inhibiting the activation of Th1 and Th17 cells that produce pro-inflammatory cytokines, thereby regulating the hyperplasia of epidermis induced by Th1/Th17 related cytokines.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory dermatosis induced by altered interactions between the immune system and skin and characterized by hyperplasia of the epidermis (acanthosis), infiltration of leukocytes into both the dermis and epidermis, and dilation and growth of blood vessels. Our previous studies have shown that topical application of indigo naturalis significantly improves psoriatic symptoms and demonstrated that the anti-psoriatic effects of indigo naturalis are mediated by promoting differentiation and inhibiting proliferation of epidermal keratinocytes. However, the potential effect of indigo naturalis on the immune system is unknown.

Currently, growing evidence demonstrates that activated T cells are the primary modulators in the pathogenesis of psoriasis and psoriasis is believed to be a mixed Th1/Th17 disease with strong IL-17 and interferon-γ (IFN-γ) signatures. The identification of elevated levels of IFN-γ, tumor necrosis factor (TNF-α), IL-12, IL-17 and IL 22 in cutaneous lesions and in the serum of psoriatic patients supports the theory that these Th1/Th17-related cytokines directly or indirectly act on keratinocytes leading to their activation and hyperproliferation. The investigators suppose the therapeutic effect of indigo naturalis in psoriasis may involve inhibiting the activation of Th1 and Th17 cells that produce pro-inflammatory cytokines, thereby regulating the hyperplasia of epidermis induced by Th1/Th17 related cytokines.

The aim of this study is:

1. To investigate whether the effect of indigo naturalis in improving psoriatic symptoms is associated with the function of Th1/Th17 cells expressing IFN-γ and IL-17 in peripheral blood of patients with psoriasis before and after therapy.
2. To investigate whether the effect of indigo naturalis in improving psoriatic symptoms is associated with the production of pro-inflammatory cytokines in peripheral blood of patients with psoriasis before and after therapy.
3. To investigate whether the effect of indigo naturalis in improving psoriatic symptoms is associated with histopathological change in psoriatic lesions and whether these pathological changes are different from the change in inflammatory and immune reactions in patients with psoriasis.
4. To investigate the effects of Th1/Th17-related cytokines and immunological factors in patients with indigo naturalis treatment on epidermal keratinocytes.
5. To detect the effect of indigo naturalis on the function of releasing cytokines (IFN-γ, IL-17, and IL-23, etc.) from monocytes in patients with psoriasis.
6. To analyze the concentration of indirubin in peripheral blood and to clarify whether the effect of indigo naturalis in improving psoriatic symptoms is: (A) a systemic effect that affects the metabolism and immune system through absorption and transdermal delivery into body. (B) a direct effect on the epidermal keratinocytes alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 - 65 years, men or women
* Diagnosed as plaque-type psoriasis by the dermatologist.
* Plaque psoriasis involving <20% of the body surface area (BSA) and the psoriasis area and severity index (PASI) <20
* If of child-bearing age, negative pregnancy test at screening, agreement to continue using birth control measures approved by the investigator for the duration of the study.
* Willingness to comply with study protocol and signed informed consent form.

Exclusion Criteria:

* A history of topically or systematically sensitivity to indigo naturalis or any component in excipient.
* Systematic therapy for psoriasis within 4 weeks of baseline including Methotrexate (MTX), immunosuppressive agents (e.g. cyclosporine), retinoid (vitamin A derivatives), biologics (e.g. Etanercept, Alefacept, Infliximab), vitamin D3 analogs and phototherapy.
* Topical therapy for psoriasis within 2 weeks of baseline including tar, corticosteroid, vitamin D3 analogs, retinoid.
* Pustular or generalized erythrodermic psoriasis.
* With abnormal liver or renal function (e.g. liver cirrhosis, hepatitis B/C, renal failure, creatinine >2.0 mg/dL, AST/ALT >3 x ULN), clinically significant abnormalities in hematology, severe uncontrolled metabolic syndrome (e.g., hypertension, diabetes mellitus, metabolic arthritis, hyperthyroidism), psychiatric disease, cancer or AIDS.
* Women who are lactating, are pregnant or are planning to become pregnant.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The change of psoriasis severity compared to the change of Th1/ Th17 related cytokines from the peripheral blood | 8 weeks
  The aim of this study is to clarify the mechanism of indigo naturalis in eliminating inflammation and in regulating the immune system by way of local or systemic effect. The investigators will evaluate the clinical efficacy which includes the mean percentage change of Psoriasis Areas Severity Index (PASI) and Body Surface Area (BSA) from baseline to week 8 as compared to the change in the Th1/ Th17 related cytokines in peripheral blood.

SECONDARY OUTCOMES:
The relationship of the change in psoriasis severity and the associated change of the concentration of indirubin from the peripheral blood. | 8 weeks
  The aim of this study is to clarify the mechanism of indigo naturalis in eliminating inflammation and in regulating the immune system by way of local or systemic effect. The investigators will evaluate the clinical efficacy which includes the mean percentage change of Psoriasis Areas Severity Index (PASI) and Body Surface Area (BSA) from baseline to week 8 as compare to the concentration of indirubin in the peripheral blood.
The relationship of the change in psoriasis severity and the associated change in the Th1/ Th17 related cytokines from the target psoriatic lesion. | 8 weeks
  The aim of this study is to clarify the mechanism of indigo naturalis in eliminating inflammation and in regulating the immune system by way of local or systemic effect. The investigators will evaluate the clinical efficacy which includes the mean percentage change of Psoriasis Areas Severity Index (PASI) and Body Surface Area (BSA) from baseline to week 8 as compared to the local immune response (the change of the histopathology from baseline to week 8).

OTHER OUTCOMES:
The change in the level of cytokines released from Th1/Th17 on epidermal keratinocytes after indigo naturalis treatment in vitro. | 8 weeks
  The investigators will measure the effect of recombinant cytokines and cultured medium collected from peripheral blood mononuclear cells of patients pre- and post-treatment with indigo naturalis on cultured epidermal keratinocytes, and explore the effect of indigo naturalis on IFN-γ, IL-17 and IL-22 produced by activated mononuclear cells of patients with psoriasis.

CONTACTS AND LOCATIONS:
Overall Officials: YIn-Ku Lin, MD., PhD., Principal Investigator — Department Traditional Chinese Medicine, Chang Gung Memorial Hospital at Keelung
Locations (1):
- Chang Gung Medical Foundation, Chang Gung University, Taoyuan District, Taiwan